CLINICAL TRIAL: NCT01015703
Title: A Phase 1, Open-Label, Dose Escalation Study of the Safety and Tolerability of CoVaccine HT™ in Healthy Adult Volunteers
Brief Title: Open-label Safety and Tolerability Study of CoVaccine HT™ in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BTG International Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PR002-CLN-pro010
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Vaccine
Keywords: Vaccine, hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CoVaccine HT (Experimental)
  Interventions: Biological: CoVaccine HT

INTERVENTIONS:
Biological: CoVaccine HT — intramuscular injection, dose escalation

SUMMARY:
The study is being conducted to explore the safety and tolerability of CoVaccine HT in healthy male and female volunteers. In this study volunteers will receive intramuscular injections of CoVaccine HT.

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females of non child-bearing potential aged 25 to 65 years inclusive and between 19 and 35 kg/m2 body mass index (BMI)
* Generally healthy as determined by pre study medical history, physical examination, 12 lead ECG.
* Negative for hepatitis B surface antigen (HBsAg), hepatitis C antibody and human immunodeficiency virus (HIV) I and II tests at screening and rapid influenza diagnostic test at admission.

Exclusion Criteria:

* History of alcohol abuse in the last 5 years or drug abuse at any time, current significant alcohol consumption.
* Fever, active infections (such as influenza) and acute gastrointestinal symptoms following prior to first dosing
* Subjects with a previous serious reaction to a vaccine, such as angioedema or anaphylaxis

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-11; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darren Wilbraham, MB., BS, Principal Investigator — Quintiles, Inc.
Locations (1):
- Quintiles Drug Research Unit, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 mg Dose: 1 mg CoVaccine HT
- 2 mg Dose: 2 mg CoVaccine HT
- 5 mg Dose: 5 mg CoVaccine HT
- 7 mg Dose: 7 mg CoVaccine HT
- 10 mg Dose: 10 mg CoVaccine HT
Period: Overall Study
Arm/Group | 1 mg Dose | 2 mg Dose | 5 mg Dose | 7 mg Dose | 10 mg Dose
Started | 10 | 10 | 10 | 10 | 10
Completed | 8 | 9 | 10 | 10 | 10
Not Completed | 2 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population, subjects who received at least one dose of test article
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 mg Dose | 2 mg Dose | 5 mg Dose | 7 mg Dose | 10 mg Dose | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (11) | 46 (11) | 49 (9) | 44 (15) | 36 (9) | 42 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 3 | 1 | 8
  Male | 9 | 8 | 9 | 7 | 9 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 2 | 4
  White | 8 | 9 | 10 | 10 | 8 | 45
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety Events
Description: Safety/tolerability study design of 5 doses of test article administered to healthy volunteers. Each dose was injected 21 days apart. Participants were withdrawn upon experiencing any adverse event.
Time Frame: Duration of study
Measure: Number; unit: percentage of patients
Arm/Group | 1 mg Dose | 2 mg Dose | 5 mg Dose | 7 mg Dose | 10 mg Dose
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
percentage of patients | 20 | 0 | 40 | 50 | 40

ADVERSE EVENTS:
Arm/Group | 1 mg Dose | 2 mg Dose | 5 mg Dose | 7 mg Dose | 10 mg Dose
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 2/10 | 0/10 | 4/10 | 5/10 | 4/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 mg Dose (N=10) | 2 mg Dose (N=10) | 5 mg Dose (N=10) | 7 mg Dose (N=10) | 10 mg Dose (N=10)
influenza-like illness (General disorders) | 2 (2) | 0 (0) | 4 (4) | 3 (3) | 4 (4)
injection site pain (General disorders) | 2 (4) | 0 (0) | 4 (5) | 5 (5) | 4 (4)
malaise (General disorders) | 2 (2) | 0 (0) | 4 (4) | 5 (5) | 1 (1)
myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 5 (5) | 1 (1)
headache (Nervous system disorders) | 2 (2) | 0 (0) | 4 (4) | 5 (5) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No